CLINICAL TRIAL: NCT03935906
Title: Reaching mEthadone Users Attending Community pHarmacies With HCV
Acronym: REACH HCV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Public Health Wales (Other Government); Burnet Institute (Other)
Responsible Party: Principal Investigator, John Dillon, Professor of Hepatology and Gastroenterology, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-025-18
Record Dates: First submitted 2019-04-15; First posted 2019-05-02 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Hepatitis C
Keywords: Point of Care; Direct Acting Antivirals; Community Pharmacy; Opiate Substitution Therapy
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reach Pathway (Experimental): Community pharmacist will explain the risks of contracting HCV from current or historical intravenous drug use. OST patients will then meet with an outreach hepatology nurse specialist who will perform a diagnostic point-of-care (PoC) HCV test along with venepuncture for safety blood tests and confirmatory HCV RNA on the pharmacy premises. The nurse will return for a subsequent visit to prescribe (in the UK; in Australia prescribing is undertaken by qualified medic) and deliver HCV medication for participants who test positive, which will be dispensed alongside their OST schedule by their community pharmacist. The outreach nurse will return after approximately 14 days to confirm negative results, dispense medication for new patients with positive results (PCR positive but below limit of detection of POC test) and confirm follow up appointments where required. The RNA and PoC test will also be administered for sustained viral response at 12 weeks post treatment (SVR12).
  Interventions: Other: Reach Pathway
- Education-only Pathway (Experimental): The community pharmacist will discuss the risks of contracting HCV through current or historical intravenous drug use. The community pharmacist will then advise participants on the nearest centre for HCV testing and treatment, as is standard of care for the countries included in this study. If they are referred from a REACH pharmacy, they will present a reply slip and/or the Patient Information Sheet to the nurse who will then consent the participant, perform HCV and safety blood tests, and complete the study paperwork. The participant's medication will be delivered to, and dispensed from, their community pharmacy alongside their OST. Participants will return to the local BBV clinic for an SVR12 test after completing treatment.
  Interventions: Other: Education-only Pathway

INTERVENTIONS:
Other: Reach Pathway — Trial of outreach nurse offering point-of-care Hepatitis C (HCV) testing to opiate substitution therapy patients in community pharmacies, which is hypothesised to improve number of patients tested and cured of HCV.
  Arms: Reach Pathway
Other: Education-only Pathway — Trial of community pharmacists advising opiate substitution therapy patients to attend a local blood-borne virus clinic to be tested for Hepatitis C by a specialist nurse, which represents the standard care pathway for HCV patients in the countries included in the study.
  Arms: Education-only Pathway

SUMMARY:
Hepatitis C Virus (HCV) is a blood-borne virus that damages the liver and is a major public health threat globally. Most individuals infected with HCV are unaware of it and show no symptoms until presenting with incurable, fatal end-stage disease. In Scotland and Australia approximately 0.7% of the general population has chronic HCV with 0.4% in Wales, and they are at risk of developing cirrhosis and hepatocellular carcinoma. The clinical challenge is to identify those infected and bring them into treatment before the disease advances.

The greatest risk factor for acquiring HCV in many countries is through injecting drug use. On the road to recovery from drug use, many will receive long-term opiate substitution therapy (OST), commonly with methadone or buprenorphine. Internationally, OST is routinely dispensed by a community pharmacist. HCV testing can be offered by GPs, drugs workers, drug agencies, social workers, community pharmacies and needle exchange sites. Once patients are diagnosed, they are referred to a hospital-based service to receive anti-HCV treatment. In this pathway, less than 10% of the OST population is tested per year, and cumulative rates of testing are less than 50% of those on OST.

Highly effective Directly Acting Antiviral (DAA) treatment combinations are now available and achieve HCV cure rates in excess of 95%, with once or twice daily tablets for 8-24 weeks.

The REACH HCV study will compare efficacy of an education-only HCV referral and treatment pathway against a nurse-led point-of-care device testing and treatment pathway among OST patients in community pharmacies in Scotland, Wales and Australia. Eligible participants will be treated using DAAs.

DETAILED DESCRIPTION:
The REACH HCV study is an international, cluster-randomised non-clinical trial with two arms. The unit of randomisation is the community pharmacy, so all participants in a given pharmacy are allocated to one of two pathways for HCV testing and treatment. There are three participating hubs located in: Scotland, Wales and Australia respectively.

The sample size is 140 participants, equally split between the three participating hubs, and the trial population is patients receiving opiate substitution therapy (OST) in community pharmacies.

Arm 1 (REACH arm): The community pharmacist will take the opportunity to explain the risks of contracting HCV from current or historical intravenous drug use. The OST patients will then meet with an outreach hepatology nurse specialist who will consent the patients and perform a diagnostic point-of-care (PoC) HCV test along with venepuncture for safety laboratory blood tests and confirmatory HCV RNA. The outreach nurse will return for a subsequent visit to prescribe (in the UK; in Australia prescribing is undertaken by qualified medic) and deliver HCV medication for those patients who test positive, which will be dispensed to participants alongside their OST schedule by their community pharmacist. The outreach nurse will return after approximately 14 days to confirm negative results, dispense medication for new patients with positive results (PCR positive but below limit of detection of POC test) and confirm follow up appointments where required. The RNA and PoC test will also be administered for sustained viral response at 12 weeks post treatment (SVR12).

Arm 2 (Education-only arm): The community pharmacist will discuss the risks of contracting HCV through current or historical intravenous drug use. The community pharmacist will then advise participants on the nearest centre for HCV testing and treatment, as is standard of care for the countries included in this study. If they are referred from a REACH pharmacy, they will present a reply slip and/or the Patient Information Sheet to the nurse who will then consent the participant, perform HCV and safety blood tests, and complete the study paperwork. The participant's medication will be delivered to, and dispensed from, their community pharmacy alongside their OST. Participants will return to the local BBV clinic for an SVR12 test after completing treatment.

All eligible HCV-infected participants will receive treatment with 100mg glecaprevir/40mg pibrentasvir (Maviret) a pan-genotypic Direct Acting Antiviral (DAA) for between 8-16 weeks, depending on blood test results. The study is planned to run for a total of two years, with one year clinical phase and one year follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Previous or current injecting drug user.
* Stable OST dose for greater than 12 weeks prior to study enrolment.
* Glecaprevir/pibrentasvir treatment naïve.
* Able to voluntarily sign and date an informed consent form prior to initiation of any screening or study specific procedures.
* Able to understand and adhere to study visit schedule and all other protocol requirements.

Exclusion Criteria:

* Female who is pregnant, planning to become pregnant or breastfeeding or unwilling/unable to take appropriate birth control.
* Known current HIV infection.
* Known current HBV infection. Serological: patients with a positive HBsAg or isolated positive anti-HBC will be excluded from the study and followed up in secondary care.
* Previous treatment with glecaprevir/pibrentasvir.
* Currently taking any concomitant medication that has a warning of'do not co-administer' with glecaprevir and/or pibrentasvir as defined by the Liverpool Hep drug interactions website and product SmPC.
* Clinically significant abnormalities that make candidate unsuitable for this study in the opinion of the investigator including but not limited to:
* Uncontrolled cardiac, respiratory, gastrointestinal, hematologic, neurologic, psychiatric or other medical disease or disorder, which is unrelated to existing HCV infection.
* History of either current or previous decompensated liver disease or symptoms/signs of decompensation e.g. ascites noted on physical exam, use of beta-blockers for portal hypertension, hepatic encephalopathy or oesophageal variceal bleeding.
* Candidate is deemed unsuitable to receive study drugs by the study investigator, for any reason according to clinical judgement.
* Unable or unwilling to provide informed consent.
* History of severe, life-threatening or other significant sensitivity to any excipients of the study drugs.
* Drug-drug Interaction which may have safety concerns with any concomitant medication the patient is receiving including non-prescribed and/or recreational drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
SVR12 | 12 weeks after participants finish their hepatitis C treatment regimen
  Proportion of patients in a population of stable opiate substitution therapy patients achieving Sustained Viral Response at 12 weeks post-treatment in the REACH pathway versus education-only pathway (Intention to Treat analysis).

SECONDARY OUTCOMES:
Determine whether the REACH pathway compared with the education only pathway leads to more people on opiate substitution therapy who are confirmed HCV RNA positive being treated and cured. | 12 weeks after participants finish their hepatitis C treatment regimen
  Percentage of patients achieving Sustained Viral Response at 12 weeks post-treatment from the patient population that tested positive for HCV in each arm (modified Intention to Treat analysis).
Cost-effectiveness analysis of the REACH pathway versus the education-only pathway, from the perspective of the NHS (UK) and Medicare (Australia). | 2 years
  Incremental cost-effectiveness ratio to consider the epidemiological impact of scaling up the intervention to all pharmacies in a specific setting in Australia, Scotland and Wales; and cost-benefit calculations (e.g. cost per HCV diagnosis; cost per SVR12; cost per HCV infection averted; number needed to screen).
Determine whether the REACH pathway compared with the education-only pathway leads to more people on opiate substitution therapy being tested for HCV. | 2 years
  Proportion of patients being tested for HCV in each arm
Compare adherence and persistence to HCV therapy in the Reach pathway to the education-only pathway. | 2 years
  Proportion of patients adhering to therapy in each arm (taking ≥ 85% of prescribed tablets) as reported in the observed therapy adherence log.
Assess the impact of baseline blood tests on treatment decisions. | 2 years
  Proportion of patients in whom changes in therapy are advised due to blood test results, as recorded at start of HCV therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Healy, PhD, Principal Investigator — Public Health Wales; Joseph Doyle, PhD, Principal Investigator — Macfarlane Burnet Institute for Medical Research and Public Health; John F Dillon, PhD, Study Director — University of Dundee
Locations (3):
- The Burnet Institute, Melbourne, Australia
- United Kingdom (2):
  - NHS Tayside, Dundee, Scotland
  - Public Health Wales, Cardiff, Wales

IPD SHARING:
Plan to Share IPD: Yes
Anonymised Individual Participant Data (IPD) will be retained by the study team. Access to IPD will be granted to researchers who supply a methodologically sound proposal. Access will be granted in line with prevailing recommendations via a reputable online controlled access repository. Requests for data access should be sent to the corresponding author (ORCID: 0000-0002-7586-7712). Data which may be shared include all IPD collected during the trial which underlie the final published results, after de-identification; the study protocol; the SAP; the Data Management Plan (DMP).
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Post-publication of final results for a period of 3 years.
Access Criteria: Researchers who supply a methodologically sound proposal.

REFERENCES:
- [Derived] Byrne CJ, Radley A, Inglis SK, Beer L, Palmer N, Duc Pham M, Allardice K, Wang H, Robinson E, Hermansson M, Semizarov D, Healy B, Doyle JS, Dillon JF. Reaching people receiving opioid agonist therapy at community pharmacies with hepatitis C virus: an international randomised controlled trial. Aliment Pharmacol Ther. 2022 Jun;55(12):1512-1523. doi: 10.1111/apt.16953. Epub 2022 May 10. PMID 35538396
- [Derived] Byrne C, Radley A, Inglis SK, Beer LJZ, Palmer N, Pham MD, Healy B, Doyle JS, Donnan P, Dillon JF. Reaching mEthadone users Attending Community pHarmacies with HCV: an international cluster randomised controlled trial protocol (REACH HCV). BMJ Open. 2020 Aug 30;10(8):e036501. doi: 10.1136/bmjopen-2019-036501. PMID 32868356